CLINICAL TRIAL: NCT04297332
Title: Promising Methods to Decrease Delay Discounting and Reduce Relapse to Smoking
Brief Title: Episodic Future Thinking and Future Thinking Priming for Smoking Cessation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: I 82819; NCI-2020-00697 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 82819 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2020-02-28; First posted 2020-03-05 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Tobacco-Related Carcinoma
MeSH Terms: interventions — Behavior Therapy; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm I (active EFT, active FTP) (Experimental): Participants are provided with Forever Free relapse prevention booklets and receive a 2-week supply of nicotine patches, gum, or lozenges. Participants also receive 1 proactive coaching call within 24 hours of quit date. Beginning on the quit date, participants complete an active episodic future thinking or active future thinking priming task once per week for 12 weeks, alternating every week between tasks.
  Interventions: Behavioral: Behavioral Intervention; Other: Informational Intervention; Other: Telephone-Based Intervention
- Arm II (active EFT, control FTP) (Experimental): Participants are provided with Forever Free relapse prevention booklets and receive a 2-week supply of nicotine patches, gum, or lozenges. Participants also receive 1 proactive coaching call within 24 hours of quit date. Beginning on the quit date, participants complete an active episodic future thinking or control future thinking priming task once per week for 12 weeks, alternating every week between tasks.
  Interventions: Behavioral: Behavioral Intervention; Other: Informational Intervention; Drug: Nicotine Replacement; Other: Telephone-Based Intervention
- Arm III (control EFT, active FTP) (Experimental): Participants are provided with Forever Free relapse prevention booklets and receive a 2-week supply of nicotine patches, gum, or lozenges. Participants also receive 1 proactive coaching call within 24 hours of quit date. Beginning on the quit date, participants complete a control episodic future thinking or active future thinking priming task once per week for 12 weeks, alternating every week between tasks.
  Interventions: Behavioral: Behavioral Intervention; Other: Informational Intervention; Drug: Nicotine Replacement; Other: Telephone-Based Intervention
- Arm IV (control EFT, control TFP) (Active Comparator): Participants are provided with Forever Free relapse prevention booklets and receive a 2-week supply of nicotine patches, gum, or lozenges. Participants also receive 1 proactive coaching call within 24 hours of quit date. Beginning on the quit date, participants complete a control episodic future thinking or control future thinking priming tasks once per week for 12 weeks, alternating every week between tasks.
  Interventions: Behavioral: Behavioral Intervention; Other: Informational Intervention; Drug: Nicotine Replacement; Other: Telephone-Based Intervention

INTERVENTIONS:
Behavioral: Behavioral Intervention — Complete active episodic thinking task
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (active EFT, active FTP); Arm II (active EFT, control FTP)
Behavioral: Behavioral Intervention — Complete active future thinking priming task
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (active EFT, active FTP); Arm III (control EFT, active FTP)
Behavioral: Behavioral Intervention — Complete control episodic future thinking task
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Arm III (control EFT, active FTP); Arm IV (control EFT, control TFP)
Behavioral: Behavioral Intervention — Complete control future thinking priming task
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Arm II (active EFT, control FTP); Arm IV (control EFT, control TFP)
Other: Informational Intervention — Provided with Forever Free relapse prevention booklet
Drug: Nicotine Replacement — Receive nicotine patches, gum, or lozenges
  Other Names: nicotine replacement therapy; NRT
  Arms: Arm II (active EFT, control FTP); Arm III (control EFT, active FTP); Arm IV (control EFT, control TFP)
Other: Telephone-Based Intervention — Receive coaching call

SUMMARY:
This trial studies the main and interactive effects of episodic future thinking and future thinking priming tasks on helping participants to quit smoking. Episodic future thinking and future thinking priming tasks may decrease delay discounting rates and reduce relapse to smoking and help participants quit smoking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To quantify the main and interactive effects of the episodic future thinking (EFT) and future thinking priming (FTP) tasks on delay discounting rate, latency to relapse, and multiple abstinence and self-regulation measures among smokers (n=76) who call a busy Quitline to quit smoking.

OUTLINE: Participants are randomized to 1 of 4 arms.

ARM I: Participants are provided with Forever Free relapse prevention booklets and receive a 2-week supply of nicotine patches, gum, or lozenges. Participants also receive 1 proactive coaching call within 24 hours of quit date. Beginning on the quit date, participants complete an active episodic future thinking or active future thinking priming task once per week for 12 weeks, alternating every week between tasks.

ARM II: Participants are provided with Forever Free relapse prevention booklets and receive a 2-week supply of nicotine patches, gum, or lozenges. Participants also receive 1 proactive coaching call within 24 hours of quit date. Beginning on the quit date, participants complete an active episodic future thinking or control future thinking priming task once per week for 12 weeks, alternating every week between tasks.

ARM III: Participants are provided with Forever Free relapse prevention booklets and receive a 2-week supply of nicotine patches, gum, or lozenges. Participants also receive 1 proactive coaching call within 24 hours of quit date. Beginning on the quit date, participants complete a control episodic future thinking or active future thinking priming task once per week for 12 weeks, alternating every week between tasks.

ARM IV: Participants are provided with Forever Free relapse prevention booklets and receive a 2-week supply of nicotine patches, gum, or lozenges. Participants also receive 1 proactive coaching call within 24 hours of quit date. Beginning on the quit date, participants complete a control episodic future thinking or control future thinking priming tasks once per week for 12 weeks, alternating every week between tasks.

ELIGIBILITY:
Inclusion Criteria:

* Smoke >= 8 cigarettes daily
* Planning to quit in the next 14 days
* No regular use of other tobacco products
* Access to the internet
* In possession of a smartphone with text messaging capabilities
* In possession of an email address accessible at least every other day

Exclusion Criteria:

* Unable or unwilling to provide consent
* Unable to provide data to the research team after the quit date
* Current use of bupropion or varenicline
* Drinking >= 20 alcoholic drinks per week
* Use of drugs of abuse in the past 30 days
* Living in the same household as a participant already enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Change in Delay discounting rate | Baseline, and 4 and 12 weeks after quit date
  Assessed with the 5-Trial Adjusting Delay Discounting.
Latency to relapse | Baseline, assessed up to 12 weeks
  Will be assessed with the Timeline Follow-Back procedure administered by telephone. Analyzed using generalized mixed models.

SECONDARY OUTCOMES:
Latency to first relapse | up to 12 weeks
  Defined as the number of days until first relapse (any smoking for seven consecutive days). Will be assessed with the Timeline Follow-Back procedure administered by telephone. Analyzed using generalized mixed models.
Number of days abstinent | Up to 12 weeks
  Will be evaluated by cox proportional-hazards survival model analyses.
7-day point prevalence abstinence rates | At 4 and 12 weeks after quit date
  Will be evaluated by cox proportional-hazards survival model analyses.
Attentional, motor, and non-planning impulsiveness | Up to 12 weeks
  Assessed with the Barratt Impulsiveness Scale.
Behavioral inhibition and behavioral activation | Up to 12 weeks
  Assessed with the Behavioral Avoidance/Inhibition scales.
Self-control | Up to 12 weeks
  Assessed with the Brief Self-Control Survey.
Ability to regulate behavior to achieve goals | Up to 12 weeks
  Assessed with the Short Self-Regulation Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Sheffer, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States